CLINICAL TRIAL: NCT01701115
Title: Effect of Local Anesthetic Dose on Interscalene Block for Shoulder Arthroscopy, Patient Satisfaction and Return of Handgrip Strength
Brief Title: Effect of Local Anesthetic Dose on Interscalene Block
Acronym: Low Dose ISB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-011
Record Dates: First submitted 2012-09-24; First posted 2012-10-04 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Arthroscopy; Interscalene Block
Keywords: Interscalene Block
MeSH Terms: interventions — Anesthetics, Local; Mepivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (20 mL) Local Anesthetic (Experimental): Intervention to be administered is a total volume of 20 mL local anesthetic containing a 1:1 mixture of 1.5% Mepivacaine: 0.5% Bupivacaine.
  Interventions: Procedure: Low Dose (20 ml) Local Anesthetic Volume for Interscalene Block; Drug: Low Dose (20 mL) Local Anesthetic (Mepivacaine:Bupivacaine)
- Control Dose (40 mL) Local Anesthetic (Active Comparator): Intervention to be administered is a total volume of 40 mL local anesthetic containing a 1:1 mixture of 1.5% Mepivacaine: 0.5% Bupivacaine
  Interventions: Procedure: Control Dose (40 mL) Local Anesthetic Volume for Interscalene Block; Drug: Control Dose (40 mL) Local Anesthetic (Mepivacaine:Bupivacaine)

INTERVENTIONS:
Procedure: Low Dose (20 ml) Local Anesthetic Volume for Interscalene Block — Anesthetic volume:
  Investigational group: A 1:1 Mepivacaine 1.5%: Bupivacaine 0.5% mixture for a total of 20 mL
  Arms: Low Dose (20 mL) Local Anesthetic
Procedure: Control Dose (40 mL) Local Anesthetic Volume for Interscalene Block — Anesthetic volume:
  Control group: A 1:1 Mepivacaine 1.5%: Bupivacaine 0.5% mixture for a total of 40 mL
  Arms: Control Dose (40 mL) Local Anesthetic
Drug: Low Dose (20 mL) Local Anesthetic (Mepivacaine:Bupivacaine)
  Other Names: Mepivacaine; Bupivacaine
  Arms: Low Dose (20 mL) Local Anesthetic
Drug: Control Dose (40 mL) Local Anesthetic (Mepivacaine:Bupivacaine)
  Other Names: Mepivacaine; Bupivacaine
  Arms: Control Dose (40 mL) Local Anesthetic

SUMMARY:
The purpose of this study is to determine if a decrease in the standard volume of local anesthetic used to numb your shoulder area before shoulder arthroscopy will provide adequate anesthesia for the procedure and decrease the amount of time until you are ready for discharge from the hospital.

DETAILED DESCRIPTION:
Traditionally, an interscalene block is done either with nerve stimulator or ultrasound guided using 40-60mL of local anesthetic. The study plans to investigate the difference in hand grip strength post-operatively in patients who will receive interscalene blocks with 40mL versus a lower dose (20mL) of local anesthetic. We suspect the lower dose will achieve adequate surgical anesthesia while creating less motor block and thus, increase patient satisfaction, present fewer complications or adverse affects and decrease time in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 80 years old
* Surgical time < 2.5 hours
* ASA I, II or III
* Shoulder arthroscopy

Exclusion Criteria:

* Age < 18 or > 80 years old
* Chronic pain patients (on narcotics/opioids > 3 months)
* Open shoulder surgical procedure
* BMI > 40
* Pre-existing neurological condition
* Patient refusal of interscalene block
* Severe respiratory disease or hemidiaphragmatic dysfunction
* Allergy to any local anesthetics
* Planned general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose (20 mL) Local Anesthetic: Intervention to be administered is a total volume of 20 mL local anesthetic containing a 1:1 mixture of 1.5% Mepivacaine: 0.5% Bupivacaine.
  Low Dose (20 ml) Local Anesthetic Volume for Interscalene Block: Anesthetic volume:
  Investigational group: A 1:1 Mepivacaine 1.5%: Bupivacaine 0.5% mixture for a total of 20 mL
  Low Dose (20 mL) Local Anesthetic (Mepivacaine:Bupivacaine)
- Control Dose (40 mL) Local Anesthetic: Intervention to be administered is a total volume of 40 mL local anesthetic containing a 1:1 mixture of 1.5% Mepivacaine: 0.5% Bupivacaine
  Control Dose (40 mL) Local Anesthetic Volume for Interscalene Block: Anesthetic volume:
  Control group: A 1:1 Mepivacaine 1.5%: Bupivacaine 0.5% mixture for a total of 40 mL
  Control Dose (40 mL) Local Anesthetic (Mepivacaine:Bupivacaine)
Period: Overall Study
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Started | 77 | 77
Completed | 75 | 77
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.5) | 50 (14.3) | 50.6 (14.1)
Sex/Gender, Customized [Number; unit: Percentage of participants]
  Female | 25.3 | 26 | 25.7
  Male | 74.7 | 74 | 74.3
Region of Enrollment [Number; unit: participants]
  United States | 75 | 77 | 152
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.2) | 26.3 (3.7) | 26.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Handgrip Strength
Description: The primary outcome will be handgrip strength as measured by a dynamometer. A reading will be obtained at baseline (before the interscalene block) and 60 minutes post-operative.
Time Frame: Difference between between baseline and postoperative.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Number analyzed (Participants) | 75 | 77
kg | 6.45 (1.6) | 2.98 (1.7)

2. Secondary Outcome: Patient Readiness to Discharge
Time Frame: Participants will be followed every 15 minutes post-surgery until discharged from the hospital (up to 180 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Number analyzed (Participants) | 75 | 77
minutes | 60 (5) | 65 (7)

3. Secondary Outcome: Duration of Analgesia
Description: Time to pain
Time Frame: Postoperative Day 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Number analyzed (Participants) | 49 | 43
minutes | 993 [635 to 1119] | 960 [759 to 1340]

4. Secondary Outcome: Side Effects
Description: Incidence of nausea
Time Frame: Postoperative Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Number analyzed (Participants) | 57 | 55
Participants | 23 | 22

ADVERSE EVENTS:
Arm/Group | Low Dose (20 mL) Local Anesthetic | Control Dose (40 mL) Local Anesthetic
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/77
Other Adverse Events (participants affected / at risk) | 0/75 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes